CLINICAL TRIAL: NCT06565793
Title: The Impact of Radiation Delivered to the Patient and the Amount of Iodinated Contrast Medium Injected in Complex Versus Noncomplex Percutaneous Coronary Intervention.
Brief Title: A MAajor RAdiation-based PCI Study in STEMI and NSTEMI
Acronym: MARAA
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Cardiologique du Nord (Other)
Collaborators: Clinica Mediterranea (Other)
Responsible Party: Principal Investigator, Francesco Nappi, Consultan, Centre Cardiologique du Nord
Other Study IDs: ID: CN-08-24
Record Dates: First submitted 2024-08-11; First posted 2024-08-22 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Myocardial Infarction (MI); Radiation Toxicity; Coronary Stenosis; Coronary Thrombosis; Coronary Artery Calcification; Coronary Occlusion; Coronary Syndrome; Coronary Artery Disease
Keywords: PCI,DES, Radiation
MeSH Terms: conditions — Myocardial Infarction; Radiation Injuries; Coronary Stenosis; Coronary Thrombosis; Coronary Occlusion; Angina, Unstable; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Non Complex PCI: The objective of this study is to examine the efficacy of percutaneous coronary intervention (PCI) with the use of drug-eluting stents (DES) in patients diagnosed with ST-Elevation Myocardial Infarction (STEMI) or Non-ST-Elevation Myocardial Infarction (NSTEMI).
  Interventions: Device: Non Complex PCI
- Complex PCI: This study focuses on patients diagnosed with either STEMI or NSTEMI who have undergone complex percutaneous coronary intervention (PCI) with the use of drug-eluting stents (DES).The following criteria were used to distinguish between complex and very complex angioplasty cases:
  The following procedures have been identified as complex or very complex:
  * Unprotected Left Coronary Common Trunk Angioplasty (UT-PCI)
  * Angioplasty with Rotablator Rotary Atherectomy (ARota-PCI)
  * Angioplasty of Chronic Coronary Occlusion (CCO-PCI)
  Interventions: Device: Complex PCI

INTERVENTIONS:
Device: Non Complex PCI — The patient cohort included individuals who had been hospitalized with a diagnosis of either STEMI or non-STEMI. The procedure involved percutaneous coronary intervention (PCI) with the use of drug-eluting stents (DES).
  Groups: Non Complex PCI
Device: Complex PCI — The patient cohort included individuals who had been hospitalized with a diagnosis of either STEMI or non-STEMI. The procedure involved complex percutaneous coronary intervention (PCI) with the use of drug-eluting stents (DES).This designation is applied to angioplasty procedures that meet at least one criterion for complexity. The complex angioplasty involved patients with unprotected left coronary common trunk (UT-PCI), the use of rotablator rotary atherectomy (ARota-PCI), the angioplasty of chronic coronary occlusion (CCO-PCI), or the angioplasty of a bifurcation lesion (CBL-PCI).The highly intricate angioplasty procedure was conducted on patients who met at least two criteria indicative of complexity.
  Groups: Complex PCI

SUMMARY:
In France and Italy, approximately 240,000 percutaneous coronary angioplasties (PCI) are performed annually, with an increasing number of complex procedures, including those involving the left coronary common trunk, a bifurcation, chronic occlusion, or requiring Rotablator Rotary Atherectomy (ARota). The medical literature lacks sufficient data regarding several key aspects of complex angioplasty. These include the epidemiological characteristics of patients undergoing such procedures, the impact of irradiation delivered and the quantity of iodine injected on these lengthy procedures, their procedural complication rate, and in-hospital mortality.

DETAILED DESCRIPTION:
A retrospective database of the hemodynamics department of the Centre Cardiologique du Nord and Clinica Mediterranea, comprising 15,630 consecutive angioplasties performed in unselected patients between February 1, 2008, and July 7, 2018, was used to identify complex angioplasties and standard angioplasties. Two categories of complex angioplasty were identified: complex angioplasty with a single complexity criterion and very complex angioplasty with two or more complexity criteria. These complex angioplasties were then compared with standard angioplasty (angioplasty with no complexity criteria).

The following criteria were employed to delineate complex or very complex angioplasties:

* Unprotected Left Coronary Common Trunk Angioplasty (UT-PCI)
* Angioplasty with Rotablator Rotary Atherectomy (ARota-PCI)
* Angioplasty of Chronic Coronary Occlusion (CCO-PCI)
* Angioplasty of a Bifurcation Lesion (CBL-PCI)

The following definitions pertain to the classification of angioplasty procedures:

* Standard angioplasty: This encompasses angioplasty procedures that do not meet the criteria for complexity.
* Complex angioplasty: This designation is applied to angioplasty procedures that meet at least one criterion for complexity.
* Very complex angioplasty: This designation is applied to angioplasty procedures that meet at least two criteria for complexity.

ELIGIBILITY:
Inclusion Criteria:

* The patient presents with a STEMI or NSTEMI requiring either a non-complex or complex PCI.

Exclusion Criteria:

-

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Standard angioplasty: This encompasses angioplasty procedures that do not meet the criteria for complexity.
  * Complex angioplasty: This designation is applied to angioplasty procedures that meet at least one criterion for complexity.
  * Very complex angioplasty: This designation is applied to angioplasty procedures that meet at least two criteria for complexity.
Sampling Method: Probability Sample
Enrollment: 15630 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Death | 30 days
  The primary end point of the study is the rate of death
Death | 1 year
  The primary end point of the study is the rate of death
Death | 5 years
  The primary end point of the study is the rate of death
Myocardial Infarction | 30 days
  The primary end point of the study is the rate of myocardial infarction
Myocardial Infarction | 1 year
  The primary end point of the study is the rate of myocardial infarction
Myocardial Infarction | 5 years
  The primary end point of the study is the rate of myocardial infarction
Stent Thrombosis | 30 days
  The primary end point of the study is the rate of stent thrombosis
Stent Thrombosis | 1 year
  The primary end point of the study is the rate of stent thrombosis
Stent Thrombosis | 5 years
  The primary end point of the study is the rate of stent thrombosis
Acute Kidney Injury | 30 days
  The primary end point of the study is the rate of acute kidney injury
Acute Kidney Injury | 1 years
  The primary end point of the study is the rate of acute kidney injury
Coronary Obstruction Requiring Intervention | 30 days
  The primary end point of the study is the rate of coronary obstruction requiring intervention
Coronary Obstruction Requiring Intervention | 1 year
  The primary end point of the study is the rate of coronary obstruction requiring intervention
Coronary Obstruction Requiring Intervention | 5 years
  The primary end point of the study is the rate of coronary obstruction requiring intervention
Increase in Tnl and Tnt Levels | 30 days
  The primary end point of the study is the rate in increase of Tnl and Tnt levels
Increase in Tnl and Tnt Levels | 1 year
  The primary end point of the study is the rate in increase of Tnl and Tnt levels
Rehospitalization | 30 days
  The primary end point of the study is the rate of rehospitalization (coronary-related or procedure-related, including heart failure)
Rehospitalization | 1 year
  The primary end point of the study is the rate of rehospitalization (coronary-related or procedure-related, including heart failure)
Rehospitalization | 5 years
  The primary end point of the study is the rate of rehospitalization (coronary-related or procedure-related, including heart failure)

SECONDARY OUTCOMES:
Target Vessel Revascularization | 1 year
  The secondary end point of the study is the rate of target vessel revascularization
Target Vessel Revascularization | 5 years
  The secondary end point of the study is the rate of target vessel revascularization
Target Lesion Revascularization | 1 year
  The secondary end point of the study is the rate of target lesion revascularization
Target Lesion Revascularization | 5 years
  The secondary end point of the study is the rate of target lesion revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Nappi, MD, Principal Investigator — Centre Cardiologique du Nord

IPD SHARING:
Plan to Share IPD: No